CLINICAL TRIAL: NCT01009151
Title: University of Michigan Heart Failure Patient Self-Management Web Portal Pilot Study
Brief Title: Heart Failure Patient Self-Management Web Portal Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Todd M. Koelling, M.D., Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00024778
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Congestive Heart Failure
Keywords: telemonitoring; internet; home monitoring system; heart failure; self management plan; web portal
MeSH Terms: conditions — Heart Failure | interventions — Patient Portals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heart Care Self Tracker (Experimental): Web-based Home Tele-monitoring system
  Interventions: Behavioral: Heart Self Care Tracker; Behavioral: Heart Care Self Tracker

INTERVENTIONS:
Behavioral: Heart Self Care Tracker — Web-based home tele-monitoring system serving congestive heart failure patients at the University of Michigan Health System. The intervention consists of daily reporting via the Internet on parameters specified in clinical protocols, including weight, blood pressure, heart rate and heart failure symptoms. These protocols contain automated trigger mechanisms when certain values are exceeded to alert the provider and the patient for the need to take appropriate remedial action. The system provides links to educational material on heart failure and reminders for self-care measures.
  Other Names: web-based self-management system; web portal
Behavioral: Heart Care Self Tracker — Web-based Home Tele-monitoring System

SUMMARY:
The proposed pilot project is aimed at assessing the feasibility, acceptability and impact of a web-based home tele-monitoring system among congestive heart failure patients at the University of Michigan Health System. The intervention consists of daily reporting via the internet on health parameters, such as weight, blood pressure, heart rate and heart failure symptoms. In addition to symptom and data reporting, the system provides links to educational material on heart failure and reminders for self-care measures. It is designed as an inexpensive, user-friendly, and clinically effective system.

Each patient will be provided with a unique name and password, and will be instructed on how to use the self-management website.

The proposed home monitoring system study holds the potential to improve the lives of heart failure patients treated at the University of Michigan Health System by empowering them to participate actively in their care and to reduce the risk of hospitalization. As heart failure represents the most common hospital diagnosis related group (DRG)among the elderly, this study offers a significant public health benefit.

DETAILED DESCRIPTION:
The study will be based on a sample of 25 heart failure patients enrolled with the UMHS Heart Failure Program who give informed consent to participate in the study. The clinical protocols and electronic software were developed by the UMHS-CVC Heart Failure Program in collaboration with the UMHS Telemedicine Resource Center. These protocols contain automated trigger mechanisms when certain values are exceeded to alert the provider and the patient for the need to take appropriate remedial action.

The UMHS Heart Failure Disease Management Program contains a registry of more than 3000 patients with heart failure problems. Currently, a multidisciplinary nursing team maintains routine contacts with these patients through telephone calls and paper records. The program has been acknowledged for its adherence to quality of care measures, and was the first to be awarded accreditation by JCAHO for ambulatory heart failure care. Despite its relative success, patients continue to be at high risk for re-hospitalization due to worsened heart function. The proposed tele-monitoring system is expected to reduce the need for re-hospitalization and to improve health outcomes by virtue of automated daily reporting and greater patient involvement in self-management. Because of its high promise, this area of research has been receiving increased attention, but so far without definitive results. Previous research has provided evidence of reduced emergency room visits and hospitalizations, improved patient compliance with care and overall cost containment among high-risk patient populations. But the studies relied on relatively expensive systems involving specialized hardware and proprietary software. The cost of these interventions presents a limitation to the broad adoption and use of the technology. The proposed project is an attempt to ascertain the optimal method from a clinical and cost standpoint for in-home telemonitoring for this large patient population that is likely to grow with the aging of the population.

The primary end-points of this pilot are: (1) patient willingness to use the system, perceptions regarding its efficacy and effectiveness and problems encountered in its use; (2) patient adherence to heart failure-specific self care practices; (3) patient health literacy and quality of life; and (4) provider perceptions of the efficacy and effectiveness of the system and problems encountered in its use.

The findings should be helpful in refining the clinical protocols and data management algorithms and establishing a solid foundation for large-scale randomized clinical trials for obtaining the necessary evidence for wide-scale adoption of these systems in the United States and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  1. Clinical diagnosis of heart failure with NYHA II-IV symptoms, or evidence of at least one heart failure hospitalization within the past 12 months.
  2. Provider permission to approach patient for enrollment
  3. Willingness to sign informed consent

Exclusion Criteria:

* Exclusion criteria include patients who are

  1. Under the age of 19
  2. Asymptomatic heart failure
  3. Prisoners
  4. Residents of long term nursing facilities
  5. Receiving dialysis
  6. Serum creatinine ≥ 3.5 mg/dL
  7. Candidates for revascularization
  8. Candidates for valve replacement or repair
  9. With comorbidity (i.e. metastatic cancer) that is likely to lead to rehospitalization or death within a 12 month period
  10. Due to a reversible cause (i.e. hypothyroidism, anemia, etc)
  11. With pulmonary arterial hypertension that is not due to left ventricular dysfunction.
  12. Pregnant women or women of child bearing potential who are actively attempting to become pregnant or are not using an accepted form of contraception

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Patient adherence to heart failure-specific self care practices, as measured by the self-care practices score. | 12 weeks

SECONDARY OUTCOMES:
Patient satisfaction and perceptions regarding utility and acceptability of the system. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Koelling, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cardiovascular Center, Ann Arbor, Michigan, United States